CLINICAL TRIAL: NCT03932617
Title: Correlation Between Changes in End-Tidal Carbon Dioxide and Stroke Volume Variation Detected by Electrical Cardiometry as A Predictor of Fluid Volume Responsiveness in Hemodynamically Unstable Patients in the Intensive Care
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Elbaiomy Abo-elkhier, Assistant lecturer, Tanta University
Other Study IDs: 32880/01/19
Record Dates: First submitted 2019-04-28; First posted 2019-05-01 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: End Tidal Carbon Dioxide; Cardiometry; Fluid Responsiveness; Shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- fluid responders
  Interventions: Device: end tidal carbon dioxide by capnography
- fluid non responders
  Interventions: Device: end tidal carbon dioxide by capnography

INTERVENTIONS:
Device: end tidal carbon dioxide by capnography — Moreover, since PETCO2 is mainly determined by tissue CO2 production (VCO2), alveolar ventilation and CO, when stable metabolic conditions are assumed and minute ventilation is kept constant, acute changes in PETCO2 have been shown to correlate strongly with changes in CO.
  Thus, PETCO2 has been suggested as a simple economic and noninvasive alternative for continuous assessment of CO in different shock states.

SUMMARY:
This study will be conducted to assess the role of end-tidal carbon dioxide (PETCO2) monitoring to predict the fluid volume responsiveness in correlation with stroke volume variation detected by electrical cardiometry in patients with hemodynamic instability.

ELIGIBILITY:
Inclusion criteria:

* Patients who will be 18 years or older.
* Patients on mechanical ventilation in the intensive care.
* Patients developing hypotension (MABP) <65 mmHg.

Exclusion Criteria:

* Patients with organ/s failure at presentation.
* Patients with deep venous thrombosis.
* Patients with limb and pelvic fractures.
* Pregnant patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Tanta University Hospital at surgical intensive care unit (SICU).
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Assessment of sensitivity and specificity of end tidal carbon dioxide monitoring in predicting fluid responsiveness in correlation with stoke volume variation detected by cardiometry | 24 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, ElGharbiaa, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol